CLINICAL TRIAL: NCT02921555
Title: Efficacy of High-dose Corticosteroid Pulses Added to Conventional Oral Corticosteroid Course for Moderate Flares of Ulcerative Colitis.
Brief Title: Endovenous Corticosteroid Pulses in Moderate Ulcerative Colitis
Acronym: CECUM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment rate
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CECUM
Record Dates: First submitted 2016-09-22; First posted 2016-10-03 (Estimated); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis
Keywords: RCT (randomized controlled trial)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Methylprednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methylprednisolone & prednisone (Experimental): Intravenous bolus of methylprednisolone followed by a decreasing conventional course of oral prednisone
  Interventions: Drug: Methylprednisolone; Drug: Prednisone
- prednisone (Active Comparator): A decreasing conventional course of oral prednisone
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Methylprednisolone — Intravenous bolus of methylprednisolone 0.5g/day for 3 consecutive days followed by a decreasing conventional course of oral prednisone (week1; 60mg/d, w2; 50mg/d, w3;40mg/d, w4; 30mg/d, w5; 20mg/d, w6; 15mg/d, w7; 10mg/d, w8; 5 mg/d, w9; 0mg/d)
  Other Names: Urbason
  Arms: methylprednisolone & prednisone
Drug: Prednisone — Conventional course of oral prednisone (week1; 60mg/d, w2; 50mg/d, w3;40mg/d, w4; 30mg/d, w5; 20mg/d, w6; 15mg/d, w7; 10mg/d, w8; 5 mg/d, w9; 0mg/d)
  Other Names: URbason

SUMMARY:
The purpose of this study is to determine the efficacy of high-dose corticosteroid pulses added to conventional oral corticosteroid course for moderate flares of ulcerative colitis.

DETAILED DESCRIPTION:
Oral corticosteroids (CS) are the treatment of choice for moderate flares of ulcerative colitis (UC) in patients who are on 5-aminosalicylic acid (5ASA) maintenance therapy. However, the efficacy of oral CS is limited, with up to 50% of remission rate in the available randomized controlled trials (RCTs). By the other hand, uncompleted disease remission after CS use, that is, clinical but not endoscopic remission, has been associated with a higher risk of hospitalizations and need for immunomodulator or colectomy in UC. Uncontrolled data suggests that intravenous CS (IV CS) may increase the remission rate and also reduce the proportion of patients developing steroid-dependency after the index course of CS.

The hypothesis of this study is that the addition of a 3-day high-dose IV CS pulses schedule administered in the outpatient infusion unit, added to a conventional oral CS course increases the endoscopic remission rate and reduces the 1-year proportion of patients developing steroid-dependency.

This is a randomized, phase IV, open-label, multicenter, controlled study.

The planned number of patients to be included is 148, distributed in two treatment arms (with or without initial high-dose CS pulse), and stratified regarding disease onset and mesalazine use.

The main end-point will be the proportion of patients with steroid-free, clinical and endoscopic remission at 8 and 54 weeks, with no rescue therapies.

The demonstration of a higher efficacy of the proposed treatment schedule would impact on a lower requirement for conventional immunosuppressive therapy (thiopurines) and biological agents, reduced hospitalizations and surgery. Moreover, this treatment regimen allows an outpatient management of moderate flares.

Baseline characteristics will be analyzed by descriptive statistical analysis by conventional methods. Categorical variables will be compared using Mann-Whitney test and continuous variables by Student T test.

In order to evaluate the primary endpoint a Chi square test will be performed to compare the proportions of patients in both study groups that achieved clinical and endoscopic steroid-free remission at 8 weeks and is maintained without steroids or salvage therapy and with no rescue therapy up to 54 weeks.

Per protocol (PP) and intention-to-treat (IT) analysis will be made The Per Protocol analysis will include all participants who did adequately adhere to the protocol, in particular those who did received the total amount of the intervention.

Missing outcomes data will be treated as non-response imputation (NRI). The intention-to treat-analysis will only include all randomized patients in the analysis, all retained in the group to which they were allocated, except those patients with missing outcomes that did not completed treatment regimen due to SAE criteria or treatment failure.

In order to evaluate the secondary endpoints a Chi square test and a Student T test will be performed for both study groups.

Cumulative probabilities of relapse, steroid dependency and surgery will be evaluated in both groups by Kaplan-Meiery, and compared by using log-rank test.

Finally, association analysis of early clinical response, clinical and endoscopic remission at week 8 and week 8 and 54 will be performed by chi-square test and Student T test; those variables that reach a Pvalue ≤ 0.1 will be included in the logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis diagnosis by Lennard-Jones criteria
* ≥18 years
* Left or extended extent of disease
* Moderate flares of ulcerative colitis according to disease activity index (DAI)
* No maintenance therapy or 5ASA treatment
* The patient is available to understand study procedures and to sign the inform consent form
* Inform Consent Form

Exclusion Criteria:

* Previous or current thiopurines, methotrexate or biological treatment
* Administration of systemic corticoids the last 6 months
* Acute or moderate systemic infection
* Diabetes mellitus or arterial hypertension
* Pregnancy or breastfeeding
* Allergic reactions associated to corticosteroids therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugeni Domènech, MD, PhD, Principal Investigator — Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa
Locations (29):
- Spain (29):
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Althaia, xarxa assistencial universitaria de Manresa, Manresa, Barcelona
  - Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Moisès Broggi, Sant Joan Despí, Barcelona
  - Consorci Hospitalari de Terrassa, Terrassa, Barcelona
  - Hospital de Galdakao, Galdakao, Bilbao
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - hospital Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital Universitario de Ourense, Ourense, Ourense
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital De La Princesa, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Mútua de Terrassa, Terrassa
  - Hospital Clínico de Valencia, Valencia
  - Hospital Universitario General de Valencia, Valencia
  - Hospital de Manises, Valencia
  - Hospital Universitari La Fe, Valencia
  - Hospital Universitario Río Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dignass A, Lindsay JO, Sturm A, Windsor A, Colombel JF, Allez M, D'Haens G, D'Hoore A, Mantzaris G, Novacek G, Oresland T, Reinisch W, Sans M, Stange E, Vermeire S, Travis S, Van Assche G. Second European evidence-based consensus on the diagnosis and management of ulcerative colitis part 2: current management. J Crohns Colitis. 2012 Dec;6(10):991-1030. doi: 10.1016/j.crohns.2012.09.002. Epub 2012 Oct 3. No abstract available. PMID 23040451
- [Background] BARON JH, CONNELL AM, KANAGHINIS TG, LENNARD-JONES JE, JONES AF. Out-patient treatment of ulcerative colitis. Comparison between three doses of oral prednisone. Br Med J. 1962 Aug 18;2(5302):441-3. doi: 10.1136/bmj.2.5302.441. No abstract available. PMID 13865152
- [Background] Hawthorne AB, Record CO, Holdsworth CD, Giaffer MH, Burke DA, Keech ML, Hawkey CJ. Double blind trial of oral fluticasone propionate v prednisolone in the treatment of active ulcerative colitis. Gut. 1993 Jan;34(1):125-8. doi: 10.1136/gut.34.1.125. PMID 8432442
- [Background] Sood A, Midha V, Sood N, Kaushal V, Awasthi G. Methylprednisolone acetate versus oral prednisolone in moderately active ulcerative colitis. Indian J Gastroenterol. 2002 Jan-Feb;21(1):11-3. PMID 11871829
- [Background] Ardizzone S, Cassinotti A, Duca P, Mazzali C, Penati C, Manes G, Marmo R, Massari A, Molteni P, Maconi G, Porro GB. Mucosal healing predicts late outcomes after the first course of corticosteroids for newly diagnosed ulcerative colitis. Clin Gastroenterol Hepatol. 2011 Jun;9(6):483-489.e3. doi: 10.1016/j.cgh.2010.12.028. Epub 2010 Dec 31. PMID 21195796
- [Background] Elliott PR, Powell-Tuck J, Gillespie PE, Laidlow JM, Lennard-Jones JE, English J, Chakraborty J, Marks V. Prednisolone absorption in acute colitis. Gut. 1980 Jan;21(1):49-51. doi: 10.1136/gut.21.1.49. PMID 7364320
- [Background] Garcia-Planella E, Manosa M, Van Domselaar M, Gordillo J, Zabana Y, Cabre E, Lopez San Roman A, Domenech E. Long-term outcome of ulcerative colitis in patients who achieve clinical remission with a first course of corticosteroids. Dig Liver Dis. 2012 Mar;44(3):206-10. doi: 10.1016/j.dld.2011.10.004. Epub 2011 Nov 11. PMID 22079262
- [Background] Rhodes JM, Robinson R, Beales I, Pugh S, Dickinson R, Dronfield M, Speirs CJ, Wilkinson P, Wilkinson SP. Clinical trial: oral prednisolone metasulfobenzoate (Predocol) vs. oral prednisolone for active ulcerative colitis. Aliment Pharmacol Ther. 2008 Feb 1;27(3):228-40. doi: 10.1111/j.1365-2036.2007.03569.x. Epub 2007 Nov 6. PMID 17988236
- [Background] Berghouse LM, Elliott PR, Lennard-Jones JE, English J, Marks V. Plasma prednisolone levels during intravenous therapy in acute colitis. Gut. 1982 Nov;23(11):980-83. doi: 10.1136/gut.23.11.980. PMID 7129207
- [Background] Llao J, Naves JE, Ruiz-Cerulla A, Marin L, Manosa M, Rodriguez-Alonso L, Cabre E, Garcia-Planella E, Guardiola J, Domenech E. Intravenous corticosteroids in moderately active ulcerative colitis refractory to oral corticosteroids. J Crohns Colitis. 2014 Nov;8(11):1523-8. doi: 10.1016/j.crohns.2014.06.010. Epub 2014 Jul 22. PMID 25066954
- [Background] Ponticelli C, Glassock RJ, Moroni G. Induction and maintenance therapy in proliferative lupus nephritis. J Nephrol. 2010 Jan-Feb;23(1):9-16. PMID 20091481
- [Background] Oshitani N, Kamata N, Ooiso R, Kawashima D, Inagawa M, Sogawa M, Iimuro M, Jinno Y, Watanabe K, Higuchi K, Matsumoto T, Arakawa T. Outpatient treatment of moderately severe active ulcerative colitis with pulsed steroid therapy and conventional steroid therapy. Dig Dis Sci. 2003 May;48(5):1002-5. doi: 10.1023/a:1023076318751. PMID 12772803
- [Background] Sood A, Midha V, Sood N, Awasthi G. A prospective, open-label trial assessing dexamethasone pulse therapy in moderate to severe ulcerative colitis. J Clin Gastroenterol. 2002 Oct;35(4):328-31. doi: 10.1097/00004836-200210000-00009. PMID 12352296
- [Background] Nagata S, Shimizu T, Kudo T, Tomomasa T, Tajiri H, Yoden A, Kagimoto S, Tahara T, Ushijima K, Uchida K, Kobayashi A. Efficacy and safety of pulse steroid therapy in Japanese pediatric patients with ulcerative colitis: a survey of the Japanese Society for Pediatric Inflammatory Bowel Disease. Digestion. 2010;81(3):188-92. doi: 10.1159/000255379. Epub 2010 Jan 19. PMID 20090334
- [Background] Kudo T, Nagata S, Ohtani K, Fujii T, Wada M, Haruna H, Shoji H, Ohtsuka Y, Shimizu T, Yamashiro Y. Pulse steroids as induction therapy for children with ulcerative colitis. Pediatr Int. 2011 Dec;53(6):974-9. doi: 10.1111/j.1442-200X.2011.03405.x. PMID 21624004
- [Derived] Llao J, Manosa M, Martin-Arranz E, Zabana Y, Navarro-Llavat M, Teller M, Garcia-Planella E, Busquets D, Monfort D, Pineda JR, Gutierrez A, Villoria A, Menchen L, Bastida G, Garcia-Alonso FJ, Rivero M, Chaparro M, de Francisco R, Merino O, Rodriguez-Lago I, Barreiro-de Acosta M, Rodriguez-Fortunez P, Rodriguez-Jimenez C, Calafat M, Domenech E; CECUM study group of the GETECCU. Addition of pulse corticosteroids to oral prednisone in moderately active ulcerative colitis: a randomized, multicentre, open-label study by GETECCU. J Crohns Colitis. 2025 Dec 5;19(11):jjaf182. doi: 10.1093/ecco-jcc/jjaf182. PMID 41258993

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylprednisolone & Prednisone: Intravenous bolus of methylprednisolone followed by a decreasing conventional course of oral prednisone
  Methylprednisolone : Intravenous bolus of methylprednisolone 0.5g/day for 3 consecutive days followed by a decreasing conventional course of oral prednisone (week1; 60mg/d, w2; 50mg/d, w3;40mg/d, w4; 30mg/d, w5; 20mg/d, w6; 15mg/d, w7; 10mg/d, w8; 5 mg/d, w9; 0mg/d)
  Prednisone: Conventional course of oral prednisone (week1; 60mg/d, w2; 50mg/d, w3;40mg/d, w4; 30mg/d, w5; 20mg/d, w6; 15mg/d, w7; 10mg/d, w8; 5 mg/d, w9; 0mg/d)
Period: Overall Study
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Started | 36 | 39
Completed | 36 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone & Prednisone | Prednisone | Total
Number analyzed (Participants) | 36 | 39 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 47 [38 to 60] | 50 [35 to 61] | 49 [37 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 20 | 21 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not responded | 36 | 39 | 75
Region of Enrollment [Number; unit: participants]
  Spain | 36 | 39 | 75
Active smokers [Count of Participants; unit: Participants] | 2 | 1 | 3
Familial inflammatory bowel disease [Count of Participants; unit: Participants] | 5 | 4 | 9
Extensive ulcerative colitis [Count of Participants; unit: Participants] — This type of ulcerative colitis affects the entire colon. Continuous inflammation begins at the rectum and extends beyond the splenic flexure.
  Participants | 21 | 17 | 38
Oral mesalazine at inclusion [Count of Participants; unit: Participants] | 28 | 31 | 59
Number of patients with Mayo Complete score at baseline [Number; unit: participants] — This baseline measure reports the number of participants with baseline Mayo Complete scores from 6 to 10" The Mayo complete score it is composed of four parts: rectal bleeding, stool frequency, physician assessment, and endoscopy appearance evaluations. Each part is rated from 0 to 3, giving a total score of 0 to 12.
  RESULTS:
  A total score of 3 to 5 points indicates mildly active disease A total score of 6 to 10 points indicates moderately active disease A total score of 11 to 12 points indicates severely active disease.
  participants | 12 | 9 | 21
Severe endoscopic activity [Count of Participants; unit: Participants] — Endoscopic activity was assessed using the Mayo endoscopic subscore (MES); it consists of a 4-point scale from inactive (grade 0) to a severely active disease (grade 3), based on endoscopic findings.
  0= Normal or inactive disease.
  1. Mild disease (erythema, decreased vascular pattern, and mild friability).
  2. Moderate disease (marked erythema, lack of vascular pattern, friability and erosion).
  3. Severe disease (spontaneous bleeding and ulcerations).
  Participants | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopic and Clincal Remission
Description: The percentage of patients with steroid-free, endoscopic remission, with no rescue therapies.
  It has been measured by Mayo endoscopic subscore (MES). MES= 0 (no friability and granularity and intact vascular pattern). MES= 1 (mild erythema or decreased vascular pattern). MES= 2 (marked erythema, absent vascular pattern, friability, and erosions). MES= 3 (spontaneous bleeding and ulceration)
Time Frame: Change from baseline at week 8
Population: All patients participating in the study had to undergo an endoscopic assessment of at least >25cm from the anal verge at baseline and after 8 weeks.
Measure: Number; unit: participants
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
participants | 11 | 10
Statistical Analysis 1: Comparison: Methylprednisolone & Prednisone vs Prednisone; Test type: Superiority; p = 0.05, Chi-squared; Mean Difference (Final Values) = 16.2
Statistical Analysis 2: Comparison: Methylprednisolone & Prednisone vs Prednisone; Test type: Superiority; p = 0.05, Chi-squared

2. Primary Outcome: Percentage of Participants With Endoscopic and Clinical Remission
Description: The proportions of patients with steroid-free, endoscopic remission, with no rescue therapies.
  It has been measured by Mayo endoscopic subscore (MES). MES= 0 (no friability and granularity and intact vascular pattern). MES= 1 (mild erythema or decreased vascular pattern). MES= 2 (marked erythema, absent vascular pattern, friability, and erosions). MES= 3 (spontaneous bleeding and ulceration)
Time Frame: Change from baseline at week 54
Population: All patients participating in the study had to undergo an endoscopic assessment of at least >25cm from the anal verge at baseline and after 54 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
Percentage of participants | 31 | 36

3. Secondary Outcome: Percentage of Patients With Clinical Remission
Description: It was measured as a decrease in the Mayo index score from baseline of at least 3 points; and a decrease of at least 30% in the rectal bleeding variable of at least 1 point or with an absolute value of 0 or 1.
  The Mayo index score is composed of four parts: rectal bleeding, stool frequency, physician assessment, and endoscopy appearance. Each part is rated from 0 to 3, giving a total score of 0 to 12. A score of 3 to 5 points indicates mildly active disease, a score of 6 to 10 points indicates moderately active disease, and a score of 11 to 12 points indicates severely active disease.
Time Frame: Change from baseline at week 8.
Population: All patients participating in the study had to undergo a clinical assessment at baseline and after 8 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
percentage of participants | 36 [28 to 44] | 39 [31 to 47]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were collected during the study, from informed consent until the last visit.
Time Frame: 12 months
Population: Information on adverse events (AEs) were collected at all study visits via spontaneous patient reporting and patient interviews at each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
Participants | 25 | 21

5. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Serious Adverse Events (SAEs) were defined as any adverse event or adverse drug reaction that resulted in death, is life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, or caused a congenital anomaly/birth defect.
Time Frame: 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
Participants | 1 | 6

6. Secondary Outcome: Levels of C-reactive Protein
Description: Clinical assessments included the analytical laboratory test. Blood samples were taken for haematology, and C-reactive protein (mg/L) levels were measured.
Time Frame: Baseline
Population: Laboratory assessments were conducted at baseline, and blood samples were collected for C-reactive protein determination.
Measure: Least Squares Mean (Inter-Quartile Range); unit: mg/L
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
mg/L | 8 [4 to 16] | 11 [4 to 27]

7. Secondary Outcome: Levels of Serum Albumin
Description: Clinical assessments included the analytical laboratory test. Blood samples were taken for haematology, and Serum albumin determination.
Time Frame: Baseline
Population: Analytical laboratory test at baseline were performed in all participants at baseline. Blood samples were taken for haematology, and Serum albumin was determined.
Measure: Least Squares Mean (Inter-Quartile Range); unit: g/L
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
g/L | 41 [38 to 43] | 40 [36 to 45]

8. Secondary Outcome: Levels of Faecal Calprotectin
Description: Faecal samples were collected at baseline, frozen and stored at -20 Celsius degrees (ºC) for central measurement of faecal calprotectin (FC).
Time Frame: Baseline
Population: FC concentration was measured using the quantitative, chemiluminescent, sandwich immunoassay Calprotectin (LIASON® DiaSorin, Italy), with a measuring range of 5-8,000 mg/g.
Measure: Number (95% Confidence Interval); unit: mg/g
Arm/Group | Methylprednisolone & Prednisone | Prednisone
Number analyzed (Participants) | 36 | 39
mg/g | 1,230 [0,281 to 1,740] | 1,710 [0,561 to 3,330]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Clinically important AEs or adverse drug reactions were also considered serious regardless of whether they met the defined criteria and included important medical events requiring intervention to prevent one of the outcomes defined as serious.
Arm/Group | Methylprednisolone & Prednisone | Prednisone
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/36 | 6/39
Other Adverse Events (participants affected / at risk) | 25/36 | 21/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylprednisolone & Prednisone (N=36) | Prednisone (N=39)
Ulcerative colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
pyrexia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Malignant neoplasm of the ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
neurogenic tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epstein Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylprednisolone & Prednisone (N=36) | Prednisone (N=39)
hyperlipidaemia (Metabolism and nutrition disorders) | 11 (11) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) — Anaemia
Sleeplessness (Nervous system disorders) | 7 (7) | 3 (3) — sleeplessness
Excitability (Nervous system disorders) | 4 (4) | 7 (7) — Excitability
Hyperglucemia (Endocrine disorders) | 3 (3) | 3 (3) — Hyperglucemia
Headache (Nervous system disorders) | 2 (2) | 2 (2) — Headache
Arterial hypertension (Blood and lymphatic system disorders) | 1 (1) | 3 (3) — Arterial hypertension
infections (Infections and infestations) | 3 (3) | 1 (1) — infections
Heartburn (Gastrointestinal disorders) | 2 (2) | 2 (2) — Heartburn
dizziness (Vascular disorders) | 0 (0) | 3 (3) — dizziness
Hypertransaminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Hypertransaminaemia
Arthromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Arthromyalgia
Tumours (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — Tumours
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cough
Transient diplopia (Eye disorders) | 1 (1) | 0 (0) — Transient diplopia
Limb oedema (Vascular disorders) | 1 (1) | 0 (0) — Limb oedema
Hyponatraemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Hyponatraemia
Acne (Endocrine disorders) | 1 (1) | 0 (0) — Acne
Acute renal dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0) — Acute renal dysfunction

LIMITATIONS AND CAVEATS:
Early termination due to low patient recruitment rate, leading to the analysis of half of the proposed sample number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT02921555/Prot_SAP_000.pdf